CLINICAL TRIAL: NCT04255771
Title: A Prospective Randomized Controlled Trial for Postoperative Adjuvant Chemotherapy for pTanyN0M0 Upper Urinary Urothelial Carcinoma With Lymphovascular Invasion
Brief Title: A Study of Postoperative Adjuvant Chemotherapy for Upper Urinary Urothelial Carcinoma With Lymphovascular Invasion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qinghua Xia,Prof (Other Government)
Responsible Party: Sponsor-Investigator, Qinghua Xia,Prof, Deputy Director of Urology, Shandong Provincial Hospital, Shandong Provincial Hospital
Organization: Shandong Provincial Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShandongPH Urology
Record Dates: First submitted 2020-01-21; First posted 2020-02-05 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Chemotherapy Effect
MeSH Terms: interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Effect of adjuvant chemotherapy on pTanyN0M0 UTUC with LVI (Experimental): This project is to explore the effect of adjuvant chemotherapy on total tumor survival time, progression-free survival time, and recurrence-free survival time in patients with pTanyN0M0 upper urinary urothelial carcinoma with lymphatic vascular invasion (LVI) through a prospective case-control study. Therapeutic value of adjuvant chemotherapy for LVI(+) patients with pT1N0M0, pT2N0M0, and pT3-4N0M0 upper urinary urothelial carcinoma, respectively.
  Interventions: Drug: Gemcitabine
- Effect of placebo on pTanyN0M0 UTUC with lymphatic invasion (Placebo Comparator): As a control, this clinical trial also set up a placebo control group. The effect of adjuvant chemotherapy was obtained by random grouping and comparing the effects of patients in the experimental group and the control group.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Gemcitabine — Standard GC (gemcitabine and cisplatin) regimen: gemcitabine 1000-1200mg/m2 intravenous infusion on days 1 and 8, cisplatin 70mg/m2 on the second day of intravenous infusion, every 3 weeks (21-day regimen) is a cycle, A total of 3 cycles.
  Other Names: Cisplatin
  Arms: Effect of adjuvant chemotherapy on pTanyN0M0 UTUC with LVI
Drug: Placebos — Use a placebo as a comparison
  Other Names: Placebo
  Arms: Effect of placebo on pTanyN0M0 UTUC with lymphatic invasion

SUMMARY:
This project is to explore the effect of adjuvant chemotherapy on total tumor survival time, progression-free survival time, and recurrence-free survival time in patients with pTanyN0M0 upper urinary urothelial carcinoma with lymphatic vascular invasion (LVI) through a prospective case-control study.

DETAILED DESCRIPTION:
This project is to explore the effect of adjuvant chemotherapy on total tumor survival time, progression-free survival time, and recurrence-free survival time in patients with pTanyN0M0 upper urinary urothelial carcinoma with lymphatic vascular invasion (LVI) through a prospective case-control study. Therapeutic value of adjuvant chemotherapy for LVI(+) patients with pT1N0M0, pT2N0M0, and pT3-4N0M0 upper urinary urothelial carcinoma, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20-85 years;
2. ECOG score 0-1 points;
3. Patients with UTUC, undergoing radical nephrectomy, pathological staging For pTanyN0M0;
4. Patients voluntarily signed informed consent.

Exclusion Criteria:

1. Obvious cardiopulmonary dysfunction, serious diabetes and other chronic diseases;
2. Obvious chemotherapy contraindications;
3. Patients have a history of other organ malignancies;
4. Combined with tumors of other sites.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Total tumor survival time | 3 years
  Effect of postoperative adjuvant chemotherapy on total tumor survival time

SECONDARY OUTCOMES:
progression-free survival time | 3 years
  Effect of postoperative adjuvant chemotherapy on progression-free survival time

OTHER OUTCOMES:
relapse-free survival time | 3 years
  Effect of postoperative adjuvant chemotherapy on relapse-free survival time

CONTACTS AND LOCATIONS:
Overall Officials: Qinghua Xia, Prof, Study Director — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China